CLINICAL TRIAL: NCT00379210
Title: Neural Effects of Mindfulness Training on Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R21AT002761-01A1 (NIH); R21AT002761-01A1 (NIH); 10012037
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2007-11

CONDITIONS: No Condition; Focus is Neural Effects of Mindfulness Training on Attention
Keywords: Attention; ERP; event-related potentials; fMRI; functional magnetic resonance imaging; MBSR; Mindfulness Based Stress Reduction; Mindfulness Meditation Training; MMT
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Meditation training group-- received Mindfulness Based Stress Management from the Penn Program for Stress Management.
  The meditation practice initially emphasized attention to a single focus. For most concentrative exercises, this focus was the breath. The sensations of breathing were to be examined closely, and when attention wandered it was to be redirected back to the breath. In other exercises, the focus of attention was to be directed to sensations within specific body parts (body scan exercise) and sensations of walking (walking meditation). During the 5th week of classes, the mindfulness training was expanded to include some explicit training in receptive attention.
  Interventions: Behavioral: Mindfulness Meditation Training (MMT)
- 2 (Active Comparator): Nutrition education group
  An active comparison condition involving nutrition education was offered. This course matched the mindfulness course in all dimensions including course duration, homework, psychosocial support, and teacher expertise. The course was taught by a nurse who had expertise in nutrition and offered a program described in the book, Nutrition for Life by Lisa Hark.
  Interventions: Behavioral: Nutrition Education course

INTERVENTIONS:
Behavioral: Mindfulness Meditation Training (MMT) — 8-week training course in mindfulness meditation
  Other Names: MBSR, Mindfulness-Based Stress Reduction
  Arms: 1
Behavioral: Nutrition Education course — 8-week course in nutrition
  Arms: 2

SUMMARY:
The purpose of this study is to examine behavioral and neural changes resulting from Mindfulness Meditation Training (MMT), and to use this knowledge in advancing our understanding of the mechanisms of attention.

DETAILED DESCRIPTION:
Mindfulness Meditation Training (MMT) has been used successfully to decrease stress, pain, and adverse health symptoms in a varied subject population. MMT has been described as "paying attention in a particular way." Although attention is a key component of meditation, little is known about the cognitive and neural changes within the human attention system that result from MMT. In this study, we examine the effects of MMT on the human attention system using neurobehavioral measures. Here MMT comprises participation in a Mindfulness-Based-Stress-Reduction (MBSR) course, while the comparison group participates in a nutrition education course, both 8 weeks long. We compare the performance and neural activity of these groups both before and after participation in the course.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (all races and ethnicities) between 18 and 40 years old
* Women of childbearing age with a negative pregnancy test within 48 hours of scanning
* In good health
* Right-handed
* Normal or corrected-to-normal vision
* English as a first language
* Able to understand and provide signed informed consent
* No history of metal in their body or other reasons why they could not undergo an Magnetic Resonance Imaging
* No history of ischemic or hemorrhagic stroke, encephalopathy or encephalitis, minimal-cognitive impairment or dementia, movement disorder such as Parkinson's disease, head trauma causing loss of consciousness, cancer involving the central nervous system

Exclusion Criteria:

* Pregnant or breast-feeding women
* Individuals with implanted metal or electronic devices that would prevent them from MRI scanning.
* Individuals with a history of neurologic dysfunction that would prevent performance on attentional tasks including: history of transient ischemic attacks, history of cerebral infarction, history of Binswanger's disease (or a history of hypertensive encephalopathy), history of intracranial hemorrhage, history of head trauma with loss of consciousness, history of encephalitis, history of extended exposure to any known neurotoxin, history of acquired cognitive impairment, history of normal pressure hydrocephalus, history of a cancer metastatic to the central nervous system, history of Parkinson's or other basal ganglia disease, history of Guillain-Barré syndrome or chronic or relapsing polyneuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amishi P Jha, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Laboratory of Dr. Amishi Jha — http://amishi.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PI Laboratory at the University of Pennsylvania Round 1 of recruitment February 1-15, 2007 Round 2 of recruitment September 7-21, 2008
Pre-assignment Details: Participants ages and gender were matched across groups. Significant prior experience with meditation or current or past neurological disorder or metal in body (for FMRI safety) were used as exclusion criteria
Groups:
- Mindfulness Training Group: Meditation training group-- received Mindfulness Based Stress Management from the Penn Program for Stress Management
- Nutrition Education Group: Nutrition education group - received information about nutrition
Period: Overall Study
Arm/Group | Mindfulness Training Group | Nutrition Education Group
Started | 30 | 30
Completed | 20 | 23
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Training Group | Nutrition Education Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (11) | 46 (12) | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Reaction Times on the Sustained Attention to Response Task.
Description: Single digits (0-9) are flashed on the screen one by one. The number 3 is the target and all other digits are non-targets. The participant is asked to press the space bar for nontargets and withhold from pressing the space bar for the target.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Mindfulness Training Group | Nutrition Education Group
Number analyzed (Participants) | 30 | 30
milliseconds | 380 (24) | 407 (22)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Nutrition Education Group; Statistical tests are evaluated at an alpha level of 0.05 (corrected, when appropriate, for multiple comparisons). Analyses are performed on both response latency and accuracy on behavioral data. For latency analyses, mean response times for correct trials are calculated for each subject. Repeated-measures ANOVA are used for omnibus tests; paired t-tests are used for individual planned contrasts, with Bonferroni-corrected significance levels to maintain a .05 alpha level; Test type: Superiority or Other; p < 0.01, ANOVA

ADVERSE EVENTS:
Arm/Group | Mindfulness Training Group | Nutrition Education Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No